CLINICAL TRIAL: NCT02011204
Title: Noninvasive Assessment of Neuromuscular Disease Using Electrical Impedance
Brief Title: Study of Electrical Impedance Myography (EIM) in ALS
Status: Completed | Type: Observational
Sponsor: Skulpt, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2013P001505
Record Dates: First submitted 2013-12-03; First posted 2013-12-13 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Amyotrophic Lateral Sclerosis; Motor Neuron Disease; Charcot-Marie-Tooth Disease; Multiple Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease; Charcot-Marie-Tooth Disease; Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- People with ALS: People diagnosed with early ALS (possible, probable, probable-laboratory supported or definite ALS according to El Escorial criteria)
  Intervention: Electrical Impedance Myography (EIM).
  Interventions: Device: Electrical impedance myography (EIM)
- Other Neurological Diseases: People with a diagnosis of a disease that mimics ALS
  Interventions: Device: Electrical impedance myography (EIM)
- Healthy Controls: Healthy Volunteers that do not have ALS or another neurological disease that mimics ALS.
  Interventions: Device: Electrical impedance myography (EIM)

INTERVENTIONS:
Device: Electrical impedance myography (EIM) — In EIM, high-frequency alternating electrical current is applied to localized areas of muscle via surface electrodes and the consequent surface voltage patterns analyzed.
  EIM is very sensitive to the compositional and structural elements of muscle. Data from both human subjects and animal disease models, including ALS, spinal muscular atrophy (SMA), and Duchenne muscular dystrophy (DMD), show that EIM may be sensitive to a variety of pathological states. It is anticipated that EIM will thus likely be able to assist in quantifying the severity of the disease affecting various muscle groups as well as in measuring changes in the disease over time.
  Other Names: EIM1102 device

SUMMARY:
This trial is studying Electrical Impedance Myography (EIM) for measuring muscle health. The trial is studying people with Amyotrophic Lateral Sclerosis (ALS), other neuromuscular diseases, and healthy volunteers to see if the EIM device can measure disease in muscle tissue.

DETAILED DESCRIPTION:
This is a multicenter, 9-month study evaluating the effectiveness of electrical impedance myography (EIM) as a diagnostic and disease-tracking tool. In addition, the following will be studied:

1. Determine EIM device's ability to discriminate between ALS and "look-alike" non-fatal, motor-predominant syndromes;
2. Track EIM progression over time and determine the best summary EIM measure that could serve as an endpoint in future clinical trials and individual patient care; and,
3. Determine whether EIM progression is predictive of a combined outcome of survival and progression as measured by ALS Functional Rating Scale, Revised (ALSFRS-R), Hand-held Dynamometry (HHD) and Vital Capacity (VC) measures.

ELIGIBILITY:
Early ALS Inclusion Criteria:

* Sporadic or familial ALS (as defined by revised El Escorial criteria)
* Onset of weakness or spasticity due to ALS ≤ 36 months prior to the Screening/Baseline Visit.
* Slow vital capacity (SVC) ≥60% of predicted for gender, height, and age

Early ALS Exclusion Criteria:

- The presence of unstable psychiatric disease, cognitive impairment, or dementia that would impair ability of the subject to provide informed consent, or a history of active substance abuse within the prior year.

ALS Disease Mimics Inclusion Criteria:

- Diagnosis of one of the following:

a. Pure Lower Motor Neuron Disease (LMND) mimics: i. Multi-focal motor neuropathy ii. Autoimmune motor neuropathy iii. Cervical or lumbosacral radiculopathies with weakness involving more than one extremity or more than a single myotome if restricted to one extremity.

iv. Multiple peripheral mononeuropathies with clinical weakness v. Charcot-Marie-Tooth Disease vi. Any condition that produces generalized or localized weakness without concomitant sensory symptoms, including myasthenia gravis or myopathy, that the evaluating physician deems mimics ALS.

b. Pure Upper Motor Neuron Disease (UMND) mimics: i. Cervical myelopathy ii. Multiple sclerosis iii. Hereditary spastic paraparesis

ALS Disease Mimics Exclusion Criteria:

* Diagnosis of possible, probable, probable-laboratory supported, or definite ALS
* Presence of positive family history of ALS.
* The presence of unstable psychiatric disease, cognitive impairment, or dementia that would impair ability of the subject to provide informed consent, or a history of active substance abuse within the prior year.

Healthy Volunteer Inclusion Criteria:

- Absence of a known neurological disorder.

Healthy Volunteer Exclusion Criteria:

* History of ALS, myopathy, neuropathy, ALS mimic disorder or other neurodegenerative disease.
* Presence of positive family history of ALS.
* The presence of unstable psychiatric disease, cognitive impairment, or dementia that would impair ability of the subject to provide informed consent, or a history of active substance abuse within the prior year.

*Please note that this is not a complete listing on all eligibility criteria.*

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People with ALS People diagnosed with early ALS (possible, probable, probable- laboratory supported or definite ALS according to El Escorial criteria)
  Other Neurological Diseases People with a diagnosis of a disease that mimics ALS
  Healthy Controls Healthy Volunteers that do not have ALS or another neurological disease that mimics ALS.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2013-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Discrimination between Groups | Duration of the Study (9 months for Group A, one visit for Groups B and C)
  Determine EIM device's ability to discriminate between ALS and "look-alike" non-fatal, motor-predominant syndromes

SECONDARY OUTCOMES:
Tracking Progression | Duration of Study, (9 months for Group A, one visit for Groups B and C)
  Track EIM progression over time and determine the best summary EIM measure that could serve as an endpoint in future clinical trials and individual patient care
Correlation with Outcome Measures | Duration of Study (9 months for Group A, one visit for Groups B and C)
  Determine whether EIM progression is predictive of a combined outcome of survival and progression as measured by ALSFRS-R, HHD and VC.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Shefner, MD, PhD, Principal Investigator — State University of New York - Upstate Medical University
Locations (6):
- United States (6):
  - St. Joseph's Hospital & Medical Center, Phoenix, Arizona
  - University of Miami Miller School of Medicine, Miami, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Skulpt, Inc, Boston, Massachusetts
  - SUNY Upstate Medical University, Syracuse, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina